CLINICAL TRIAL: NCT00633295
Title: An Open-label, Multi-center Study to Evaluate the Efficacy and Safety of Nilotinib in Adult Patients With Gastrointestinal Stromal Tumors Resistant or Intolerant to Imatinib and or to 2nd Line Tyrosine Kinas (TK) Inhibitor
Brief Title: Phase II Study Aiming to Evaluate the Efficacy and Safety of Nilotinib Patients With Gastrointestinal Stromal Tumors (GIST) Resistant or Intolerant to Imatinib and or to 2nd Line Tyrosine Kinas (TK) Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107DIL02
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Gastrointestinal Stromal Tumors (GIST)
Keywords: GIST; TKI; IMATINIB; NILOTINIB; AMN107
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib

ARMS (1):
- nilotinib (Experimental)
  Interventions: Drug: AMN107- NILOTINIB

INTERVENTIONS:
Drug: AMN107- NILOTINIB — The dose of nilotinib will be 400 mg bid.

SUMMARY:
The mainstay of therapy for GISTs is surgical resection, however, recurrence is almost inevitable in high-risk tumors and secondary surgery or other salvage therapy has yielded poor outcome. The median survival for patients with unresectable or metastatic GIST is approximately 20 months, and for patients with local recurrence it is 9 to 12 months. Responses to chemotherapy have been at best 5%. The introduction of imatinib has dramatically changed the prognosis of these patients yielding response rates between 41% and 71% and an overall clinical benefit (tumor responses plus stable disease) ranging between 73% and 90%.

However, resistance to imatinib may develop and represents a further clinical challenge. Sunitinib has recently been approved by the FDA for patients whose disease has progressed or who are intolerant to imatinib therapy. Patients with tumor progressing on sunitinib or another 2nd line agent have limited therapeutic alternatives. Reinstitution of imatinib, if possible, is considered an acceptable option for these patients because it may slow the rate of disease progression even in the setting of prior imatinib failure; however a more optimal 3rd line treatment is needed. AMN107 is a novel aminopyrimidine, available as an oral formulation that is ATP -competitive inhibitor of BCR-ABL,more potent than Imatinib. It inhibits proliferation and autophosphorylation of 32 out of 33 BCR-ABL point mutations. In addition AMN107 also inhibits PDGFRα,PDGFRβ, and KIT. Preliminary data from an ongoing Phase I study in imatinib-resistant GIST patients (CAMN107A2103) indicate that AMN107 alone (400 mg BID) and in combination with imatinib (imatinib 400 mg BID plus AMN107 200 mg QD and 400 mg QD) is well tolerated in this pre-treated patients.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years at Visit 1
* Radiological confirmation of disease progression (CT scan PET-CT, or MRI) during imatinib therapy, on 600- 800 mg per day for at least 6 weeks.
* Radiological confirmation of disease progression (CT scan or MRI and PET-CT) during 2nd line TK inhibitor therapy.
* Patients who were intolerant to Imatinib or second line TK inhibitor (like :sunitinib). Intolerance (at any dose and/or duration), is defined as patients who did not progress on imatinib or sunitinib and have discontinued imatinib and or sunitinib therapy due to any ≥ Grade 3 adverse events that persist in spite of optimal supportive care. Patients with Grade 2 adverse events related to imatinib or sunitinib therapy, in spite of optimal supportive care measures, that persist for ≥ one month or that recurs for more than 3 times whether the dose is reduced or discontinued will also qualify patients as intolerant

Exclusion criteria:

* Prior treatment with nilotinib
* Treatment with any investigational drug ≤ 4 weeks prior to Visit 1 with the exception of imatinib and sunitinib therapy .

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of nilotinib in GIST patients resistant or intolerant to imatinib and or 2nd line TK inhibitor as measured by tumor up take of FDG PET quantitated by maximum | 6 months

SECONDARY OUTCOMES:
To assess the safety and tolerability of nilotinib as measured by rate and severity of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Litwinsky